CLINICAL TRIAL: NCT06668506
Title: A Multi-center, Prospective, Observational Study to Evaluate Improvement Effect of Subjective Symptoms of Mucotra SR Tablet in Patients With Gastritis
Brief Title: To Evaluate Improvement Effect of Subjective Symptoms of Mucotra SR Tablet in Patients With Gastritis
Status: Completed | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: MUC0S_OS_01
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mucotra® SR Tab: Mucotra® SR Tab Rebamipide 150mg

SUMMARY:
This study aims to evaluate the improvement effect on subjective symptoms of gastritis and adverse events through patient self-assessment results (PRO) by conducting follow-up observations for patients with gastritis at 2 to 4 weeks after administration of Mucotra® SR tablets.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 19 years
* Subjects with acute or chronic gastritis, requiring treatment with Mucotra® SR tab
* Subjects with subjective symptoms
* Subjects who voluntarily consent to participate in this observational study

Exclusion Criteria:

* Subjects who have had a hypersensitivity reaction to the components of Mucotra® SR tab
* Subject with genetic disorders such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The minimum number of study subjects required to estimate the two-sided 95% confidence interval of the change in the total score of subjective symptoms at 2 weeks compared to the baseline as -3.19 to 2.99, with the standard deviation assumed by referring to the AD-203P3 literature, is calculated to be 15,247 ( PASS 13. NCSS, LLC. (Kailsville, Utah, USA)
Sampling Method: Probability Sample
Enrollment: 2814 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Change in total subjective symptom score compared to baseline | 2 weeks (up to 4 weeks)
  Change in total subjective symptom score compared to baseline at 2 weeks (up to 4 weeks) on a scale of 0 to 3 points for 8 items (epigastric pain, severe pain, nausea/vomiting, acid reflux, bloating, poor appetite, heartburn, burping). Higher scores are indicative of more severe symptoms.

SECONDARY OUTCOMES:
Change in individual subjective symptom score compared to baseline | 2 weeks (maximum 4 weeks)
  Change in individual subjective symptom score compared to baseline at 2 weeks (up to 4 weeks) on a scale of 0 to 3 points for 8 items (epigastric pain, severe pain, nausea/vomiting, acid reflux, bloating, poor appetite, heartburn, burping). Higher scores are indicative of more severe symptoms.
The effective rate of subjective symptoms compared to baseline | 2 weeks (maximum 4 weeks)
  The effective rate of subjective symptoms compared to baseline at 2 weeks (maximum 4 weeks). The effective rate is the percentage of patients whose total subjective symptom scores are reduced by more than 50% compared to their scores before administration.
Overall change assessed by study subjects after administration of the study drug | 2 weeks (maximum 4 weeks)
  Overall change assessed by study subjects after administration of the study drug at 2 weeks. (maximum 4 weeks) The overall change is assessed using five criteria: very much improved, much improved, minimally improved, no change, and worse.
Overall change assessed by the researcher after administration of the drug under study | 2 weeks (maximum 4 weeks)
  Overall change assessed by the researcher after administration of the drug under study at 2 weeks (maximum 4 weeks). The overall change is assessed using five criteria: very much improved, much improved, minimally improved, no change, and worse.
Adverse events that occurred after administration of Mucotra® extended-release tablets | 2 weeks (maximum 4 weeks)
  Adverse events that occurred after administration of Mucotra® extended-release tablets at 2 weeks (maximum 4 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Song Kwang Seon Internal medicine clinic, Wŏnju, South Korea

IPD SHARING:
Plan to Share IPD: Undecided